CLINICAL TRIAL: NCT05781568
Title: Use of Blood Biomarkers for the Early Diagnosis of Hepatocellular Carcinoma (HCC)
Acronym: GALAD
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Dr. Raffaele Cozzolongo (Unknown); Dr. Palma Aurelia Iacovazzi (Unknown); Dr. Vito Giannuzzi (Unknown); Dr. Francesco Losito (Unknown); Dr. Marianna Zappimbulso (Unknown)
Responsible Party: Principal Investigator, Dr. Endrit Shahini, Principal Investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: RC202214
Record Dates: First submitted 2023-02-15; First posted 2023-03-23 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: HCC; Cirrhosis, Liver; NAFLD; HBV; HCV
Keywords: alpha fetoprotein; des-γ-carboxy-prothrombin; α-FP-L3; GALAD; GALADUS
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: The control group will be composed of patients who will be candidates for HCC surveillance, i.e. those with liver cirrhosis or chronic hepatitis of any aetiology without HCC seen at our institution.
  Included in this group are:
  1. Patients newly enrolled and who will be tested for α-FP, α-FP-L3%, and DCP as part of their regular follow-up;
  2. Patients who had previously given consent for the storage of a serum sample in the Biobank and who had authorized the dosage of α-FP, α-FP-L3% and DCP.
  Interventions: Diagnostic Test: Biomarker dosage
- Case Group: The case group will be composed of patients with newly diagnosed HCC in the context of cirrhosis or any other aetiology during the same study period. This group will include:
  1. Patients newly enrolled and who will be tested for α-FP, α-FP-L3%, and DCP as part of their regular follow-up;
  2. Patients who had previously given consent for the storage of a serum sample in the Biobank and who had authorized the dosage of α-FP, α-FP-L3% and DCP at the time of tumor diagnosis.
  Interventions: Diagnostic Test: Biomarker dosage

INTERVENTIONS:
Diagnostic Test: Biomarker dosage — The simultaneous dosage of the 3 serum biomarkers will be performed at the Clinical Pathology Laboratory, using the instrument: µTASWakoTM i30 (Micro Total Analysis System) - Fujifilm.

SUMMARY:
The objective of this observational study is to evaluate the clinical utility of the combined assay of 3 biomarkers: α-FP, α-FP-L3 and DCP (simultaneously measured by µTASWakoTM i30 automated in vitro diagnostic system) in high-risk subjects to develop this neoplasm.

In particular, it aims to:

* Evaluate the clinical utility of the combined use of α-FP, α-FP-L3 and DCP in predicting the onset of HEPATOCARCINOMA (HCC);
* Evaluate the performance of GALAD and GALADUS scores in the early diagnosis of HCC;
* Evaluate the association between the levels of the three biomarkers (individually and in combination with each other) and the stage of HCC

DETAILED DESCRIPTION:
HCC occurs in 70-95% of cases in patients with chronic liver disease, rarely in a "healthy" liver. Globally about 80% of HCCs are associated with hepatitis B virus (HBV) or hepatitis C virus (HCV) infection and their geographical distribution closely correlates with their epidemiology. Approximately 1/3 of patients with liver cirrhosis will develop HCC in the long term, with an annual risk ranging from 1%-8%.

Chronic viral hepatitis C (CHC) and chronic viral hepatitis B (CHB) together with cirrhosis of the liver respectively represent the most important risk factors in Western and Eastern Europe and therefore prolonged surveillance and prevention is recommended in these patients.

Therefore, early diagnosis of HCC is of paramount importance to prolong overall survival. Today, only about 30% of patients in Europe are diagnosed at an early stage, where curative treatments are possible.

Patients with a history of chronic liver disease are at risk of developing HCC and for this reason should undergo a screening program aimed at the early diagnosis of HCC. Asymptomatic patients but with familial predisposition on a genetic basis, according to recent international guidelines, they must be monitored periodically.

Imaging (ultrasonography, CT, and MRI), biopsy with histological examination, and blood alpha-fetoprotein measurements are used in diagnostics and staging. However, current screening/surveillance tools are not perfect.

The most popular screening tools for HCC are as follows and are performed on a semi-annual basis:

1. Abdominal ultrasound: Abdominal ultrasound is the diagnostic tool of first choice, with a sensitivity of 48% (95%CI:34-62%) and a specificity of 97% (95%CI:95-98%) as emerges from a rigorous systematic review of 14 studies of 2524 cases.
2. Tumor markers: Alpha-fetoprotein (α-FP) is a specific tumor marker. Its diagnostic sensitivity of HCC is 25-60% while its specificity is 76-96%. An α-FP level above 400 ng/mL is strongly diagnostic, but approximately two-thirds of patients with HCC <4 cm has α-FP levels <200 ng/mL and also approximately 20% of HCCs do not produce α-FP. The carbohydrate chain of α-FP is modified by fucosyltransferase during HCC development to give rise to lectin-bound α-FP (α-FP-L3) (sensitivity:40-90%; specificity:>90%) . The ratio of fucosylated α-FP to total α-FP is expressed as α-FP-L3%. Des-γ-carboxy-prothrombin (DCP or PIVKA-II) is an immature prothrombin, lacking carboxylation at various residues of glutamate (sensitivity: 48-62%; specificity: 81-98%). α-FP-L3 and DCP have been used routinely for 20 years in Japan. The combined use of these markers has increased the possibility of early detection of small HCCs. Prothrombin is formed after γ-carboxylation of vitamin K-dependent propeptides. DCP is produced due to an acquired post-translational defect in the carboxylase-vitamin K-dependent sequence of malignant cells.

   Thus, DCP production is not increased in chronic hepatitis or cirrhosis, making it a potential marker to be used in the diagnosis of HCC. However, DCP measurement has no prognostic value in cases of vitamin K deficiency or inhibition of vitamin K function (for example in subjects on TAO with dicumarols) since its synthesis is also induced by the absence of vitamin K causing false values positive. For this reason DCP is also known as PIVKA-II (protein induced in vitamin K absence). Notwithstanding these limitations, many studies have demonstrated that PIVKA-II has a high sensitivity and specificity compared to α-FP in differentiating HCC from other chronic liver diseases. Liebman et al. demonstrated that PIVKA-II can be used not only as a very specific marker for HCC but also as a prognostic factor of HCC patients. The sensitivity, specificity, and odds ratio in HCC <5 cm is 0.14-0.54, 0.95-0.99, and 6.86-29.7, respectively, with a cut-off of 40mAU /ml, and 0.07-0.56, 0.72-1 and 3.56-3 with a cut-off of 100mAU/ml. In a large study of 270 HCC patients who all had serum α-FP levels below 20 ng/mL, the combined use of the biomarkers α-FP-L3 and DCP detected 49% of all HCC patients of size less than 2cm. Furthermore, α-FP-L3 measurements with the highly sensitive method before treatment were more useful for the diagnosis and prognosis of HCC than with the conventional method. More recently, the three markers (α-FP, α-FP-L3 and DCP) showed a sensitivity and specificity of 85% (n=304 HCC patients versus 403 controls) in the early diagnosis of HCC in a German cohort.
3. Second-level investigations are CT and MRI: Useful in confirming the diagnosis and staging the disease in order to set up the correct therapeutic procedure.

"Biomarkers of HCC and their clinical significance"

Ideally, the use of serum biomarkers with adequate sensitivity and specificity could allow early diagnosis of HCC by avoiding surveillance with ultrasonography. A number of serum biomarkers, other than α-fetoprotein (α-FP) have been included in some score systems for the prediction of HCC.

However, at present, none of the biomarkers have been validated in phase III clinical trials and are used in clinical practice, except for α-FP and DCP (or PIVKAII), which are recommended by the Japanese HCC guidelines. This can be explained by the high heterogeneity of HCC biology, where alterations of different biochemical pathways are involved in the tumourigenesis process. Indeed, patients with HCC show various patterns of positivity for biomarkers of HCC.

CLINICAL STUDY DESIGN As previously indicated, this is a retrospective and prospective observational study in which the biomarkers useful for evaluating the possible progression of chronic liver disease in HCC will be dosed in two groups, a "Case" group and a "Control" group.

The need to identify biomarkers useful for predicting the possible onset of HCC in patients with chronic liver disease arises from the fact that:

1. For the majority of patients, HCC is completely asymptomatic;
2. HCCs can only be symptomatic if large;
3. α-FP tumor marker is a specific tumor marker but its diagnostic sensitivity is reduced and also about 20% of HCCs do not produce α-FP;
4. Although α-FP is being diagnosed and screened as a specific and well-established tumor marker, there is a pressing need to use highly specific and new generation biomarkers to allow an even earlier and more accurate diagnosis in patients at risk ;
5. Several studies have demonstrated that α-FP-L3 and DCP are complementary and essential markers in the early detection of HCC;
6. The combined use of α-FP, α-FP-L3 and DCP with HCC surveillance could increase the chance of detecting HCC at an early stage;
7. The combined use of these three markers would provide: Greater clinical sensitivity and effective prognostic and predictive value for early recognition of HCC;
8. The GALAD score (and GALADUS) demonstrated the efficacy of these new biomarkers in HCC prevention and surveillance programs especially in patients with liver cirrhosis almost regardless of etiology.

The following will be enrolled in the study, after signing the informed consent:

1. Patients newly diagnosed with HCC (Case group)
2. Follow-up patients with viral, NASH and/or alcoholic cirrhosis who carry out HCC prevention programs at the Gastroenterology Department I of the IRCCS "Saverio de Bellis". (control group).

The study will last for two years, and it is expected to enroll at least 30 patients for each group.

Upon enrollment and after 6 months, at follow-up, the patients belonging to both groups will have a blood sample taken to proceed with the dosage of the biomarkers.

The control group will be composed of patients who will be candidates for HCC surveillance, i.e. those with liver cirrhosis or chronic hepatitis of any aetiology without HCC seen at our institution.

Included in this group are:

1. Patients newly enrolled and who will be tested for α-FP, α-FP-L3%, and DCP as part of their regular follow-up;
2. Patients who had previously given consent for the storage of a serum sample in the Biobank and who had authorized the dosage of α-FP, α-FP-L3% and DCP.

Control patients will be required to undergo a 6-month follow-up following GALAD score evaluation to confirm the absence of HCC. These patients should have a negative multiphasic contrast-enhanced CT, MRI, or liver biopsy at the time of GALAD score evaluation.

The case group will be composed of patients with newly diagnosed HCC in the context of cirrhosis or any other aetiology during the same study period. This group will include:

1. Patients newly enrolled and who will be tested for α-FP, α-FP-L3%, and DCP as part of their regular follow-up;
2. Patients who had previously given consent for the storage of a serum sample in the Biobank and who had authorized the dosage of α-FP, α-FP-L3% and DCP at the time of tumor diagnosis.

Any patients undergoing therapy with Warfarin, an anticoagulant, will be excluded since it can increase DCP levels in the absence of HCC, risking giving false positives.

Considering that the study foresees a follow-up of at least 6 months of the recruited subjects and therefore rather long times are envisaged for its completion, it is conceivable that some patients will be lost and that the initial population will decrease. For this reason, recruitment will proceed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Case Group:

   * Patients with HCC first diagnosed from cirrhosis or other aetiology
2. Controls group:

   * Candidate patients for HCC surveillance, with liver cirrhosis and chronic hepatitis of any etiology without HCC seen at our institution

Exclusion Criteria:

* Patients treated with Warfarin, an anticoagulant, as it can increase DCP levels in the absence of HCC, risking giving false positives

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To participate in this study, patients belonging to the Gastroenterology 1 department of the IRCCS "Saverio de Bellis" will be enrolled.
  The control group will be composed of patients who will be candidates for HCC surveillance, i.e. those with liver cirrhosis or chronic hepatitis of any aetiology without HCC seen at our institution.
  The case group will be composed of patients with newly diagnosed HCC in the context of cirrhosis or any other aetiology during the same study period.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-06-27 (Estimated); Study Completion 2025-01-27 (Estimated)

PRIMARY OUTCOMES:
Biomarker dosage | six months
  Determine the GALAD alghoritm (Gender,Age, AFP-L3, AFP and Des-carboxy-prothrombin) by evaluating the values of AFP, AFP-L3, Des-carboxy-prothrombin for each patient, since the GALAD score had a high diagnostic performance as compared to each standalone markers in identifying HCC at any stage.

CONTACTS AND LOCATIONS:
Overall Officials: Endrit Shahini, MD, Principal Investigator — IRCCS "Saverio de Bellis" - Castellana Grotte (BA) - Italy
Locations (1):
- RCCS "Saverio de Bellis", Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Background] Demirtas CO, Brunetto MR. Surveillance for hepatocellular carcinoma in chronic viral hepatitis: Is it time to personalize it? World J Gastroenterol. 2021 Sep 7;27(33):5536-5554. doi: 10.3748/wjg.v27.i33.5536. PMID 34588750
- [Background] Stefaniuk P, Cianciara J, Wiercinska-Drapalo A. Present and future possibilities for early diagnosis of hepatocellular carcinoma. World J Gastroenterol. 2010 Jan 28;16(4):418-24. doi: 10.3748/wjg.v16.i4.418. PMID 20101765
- [Background] Yang JD, Addissie BD, Mara KC, Harmsen WS, Dai J, Zhang N, Wongjarupong N, Ali HM, Ali HA, Hassan FA, Lavu S, Cvinar JL, Giama NH, Moser CD, Miyabe K, Allotey LK, Algeciras-Schimnich A, Theobald JP, Ward MM, Nguyen MH, Befeler AS, Reddy KR, Schwartz M, Harnois DM, Yamada H, Srivastava S, Rinaudo JA, Gores GJ, Feng Z, Marrero JA, Roberts LR. GALAD Score for Hepatocellular Carcinoma Detection in Comparison with Liver Ultrasound and Proposal of GALADUS Score. Cancer Epidemiol Biomarkers Prev. 2019 Mar;28(3):531-538. doi: 10.1158/1055-9965.EPI-18-0281. Epub 2018 Nov 21. PMID 30464023
- See also: 10 Asks to Improve Liver Cancer Care in Europe — https://easl.eu/wp-content/uploads/2021/06/1.-EASL-Open-Letter-on-Liver-Cancer-Care.pdf